CLINICAL TRIAL: NCT06023134
Title: Clinical Characteristics and Outcomes of Patients With Pulmonary Hypertension Associated Right Heart Failure
Status: Active, not recruiting | Type: Observational
Sponsor: Jingyi Ren (Other)
Responsible Party: Sponsor-Investigator, Jingyi Ren, Professor, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Other Study IDs: PH-RHF
Record Dates: First submitted 2023-08-29; First posted 2023-09-05 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Right Heart Failure; Pulmonary Hypertension
Keywords: Right heart failure; Prognosis; Right ventricular function; Pulmonary hypertension; Biomarkers; diagnosis
MeSH Terms: conditions — Heart Failure; Hypertension, Pulmonary; Disease | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: Participants met the indication for right heart catheterization but did not meet the diagnostic criteria for pulmonary hypertension and right heart failure.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Right heart catheterization
- Pulmonary Hypertension group: Participants were classified according to the 2022 ESC/ERS guidelines for the diagnosis and treatment of pulmonary hypertension, meaning that a mean pulmonary artery pressure (mPAP) ≥20 mmHg was defined as PH.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Right heart catheterization
- Right heart failure group: Right heart failure was considered present when RV fractional area change (FAC) was <35% or tricuspid annular systolic velocity (RV S') was <9.5 cm/s or tricuspid annular plane systolic excursion (TAPSE) <17mm.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Right heart catheterization

INTERVENTIONS:
Diagnostic Test: Echocardiography — Echocardiography will be used for specific right ventricular measurements or findings: TAPSE, TAPSE:PASP ratio, tissue Doppler velocity at lateral tricuspid annulus, fractional area change, right ventricular strain, right ventricular hypertrophy, right atrial size, volumes, ejection fraction, tricuspid and pulmonary regurgitation, inferior vena cava diameter and collapsibility, shift of interventricular septum, further assisting the diagnosis of RHF.
Diagnostic Test: Right heart catheterization — Right heart catheterization is the "gold standard" for the diagnosis of PH. It also allows for direct measurement of intracardiac and pulmonary pressures, as well as cardiac output, and is commonly used to estimate right ventricular preload and afterload.

SUMMARY:
The study aims to describe the clinical characteristics and clarify the predictors of the short- and long-term outcomes of RHF patients, further assist the diagnosis, risk stratification and treatment of RHF.

DETAILED DESCRIPTION:
Right heart failure(RHF) is a clinical syndrome with symptoms, signs, and evidence of right ventricular systolic and/or diastolic dysfunction. For many years, it was largely neglected in the consideration of left-sided heart failure, while it is now evident that RHF is not only common but its presence also strongly contributes to increased morbidity and mortality. The in-hospital mortality of RHF is 7%, and the 30-day readmission rate is 20%. Therefore, diagnosis, potential treatment strategies, and prognosis improvement have become an unmet need in the field of cardiovascular disease.

In clinical practice, accurate diagnosis of RHF is the key to timely initiation of treatment and improvement of prognosis. Although current guidelines recommend clinical symptoms and signs combined with echocardiography, cardiac magnetic resonance, and other imaging means to evaluate right heart dysfunction for comprehensive diagnosis of right heart failure, the key diagnostic indicators included are inconsistent, the weight ratio of each indicator is different, the diagnostic threshold is not uniform, and the lack of comprehensive diagnostic model system brings great challenges to clinical practice.

This study aims to integrate multiple clinical biomarkers, imaging, and hemodynamic data to describe the clinical characteristics, establish noninvasive easy-to-use diagnosis models for right heart failure, and explore the risk factors for short- and long-term poor prognosis in patients with RHF.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years at the time of consent
2. Acceptation of right heart catheterization examination
3. Able to perform the entire protocol

Exclusion Criteria:

1. Life expectancy of less than 1 year based on the investigator's clinical judgment
2. Pregnant or nursing
3. Malignancy
4. Planned to undergo heart transplantation or device implantation
5. Acute coronary syndrome, uncontrolled severe arrhythmia and shock.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants who met the indications for right heart catheterization were monitored by hemodynamics and evaluated cardiac function by echocardiography. Those who met the diagnostic criteria for pulmonary hypertension were included in the pulmonary hypertension group, those who also met the diagnostic criteria for right heart failure were included in the right heart failure group, and the rest of the patients were included in the control group.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Time to first event of adjudicated CV death mortality or adjudicated HHF | 24 weeks
  The composite primary endpoint for this trial is the time to first event of adjudicated CV death or adjudicated hospitalization for heart failure （HHF） in patients with right heart failure.

SECONDARY OUTCOMES:
Occurrence of adjudicated HHF (first and recurrent) | 24 weeks
  any hospital admission due to HHF in 24 weeks
Time to adjudicated CV death | 24 weeks
  any CV death in 24 weeks
Time to all-cause mortality | 24 weeks
  any all-cause mortality in 24 weeks
Time to first all-cause hospitalisation | 24 weeks
  any hospital admission in 24 weeks
Composite of time to first event of all-cause mortality and all cause hospitalisation | 24 weeks
  The composite primary endpoint for this trial is the time to first event of all-cause mortality and all cause hospitalisation in patients with pulmonary hypertension
Change in NYHA class from baseline at week 24 | 24 weeks
  Patients are assessed for NYHA class at each admission
Changes in N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) from baseline over time | 24 weeks
  Change from baseline to week 24 in N-terminal pro-brain natriuretic peptide (NT-proBNP).Baseline value was defined as the mean of all available measurements at the time of the first right heart catheterization
Change in liver functions from baseline over time | 24 weeks
  Change of transaminase or bilirubin from baseline to week 24 .Baseline value was defined as the mean of all available measurements at the time of the first right heart catheterization
Change in renal function from baseline over time | 24 weeks
  Change of estimated Glomerular Filtration Rate from baseline to week 24. The baseline value was defined as the mean of all available measurements at the time of the first right heart catheterization
Change in echocardiographic data from baseline over time | 24 weeks
  Change from baseline to week 24 in echocardiographic data. Baseline value was defined as the mean of all available measurements at the time of the first right heart catheterization
Change in ECG data from baseline over time | 24 weeks
  Change from baseline to week 24 in ECG data.Baseline value was defined as the mean of all available measurements at the time of the first right heart catheterization

CONTACTS AND LOCATIONS:
Overall Officials: Jingyi Ren, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No